CLINICAL TRIAL: NCT00530634
Title: Multimodality Therapy for Stages II and III Non-Small Cell Lung Cancer: Surgical Resection Followed by Sequential Administration of Gemcitabine Plus Cisplatin Chemotherapy and Radiation Therapy
Brief Title: Surgery, Gemcitabine, Cisplatin, and Radiation Therapy in Treating Patients With Stage II or Stage III Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99077; P30CA033572 (NIH); CHNMC-99077; CDR0000564760 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Results first posted 2015-09-17 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Lung Cancer
Keywords: stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Gemcitabine; Gene Expression Profiling; Reverse Transcriptase Polymerase Chain Reaction; Immunohistochemistry; Chemotherapy, Adjuvant; Radiotherapy

ARMS (1):
- Gemcitabine + Cisplatin (Experimental): Surgical resection followed by (within 60 days) by chemotherapy (Gemcitabine at 1000 mg/m2 IV over 30 minutes on days 1 and 8 of a 21 day cycle and Cisplatin at 75 mg/m2 IV over 1 hour on day 8 of a 21 day cycle) followed by radiation therapy (treated using linear accelerator with photon beam energy of 6-21 MV) upon completion of 3 cycles of chemotherapy.
  Interventions: Drug: cisplatin; Drug: gemcitabine hydrochloride; Genetic: gene expression analysis; Genetic: reverse transcriptase-polymerase chain reaction; Other: immunohistochemistry staining method; Procedure: adjuvant therapy; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride
Genetic: gene expression analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: immunohistochemistry staining method
Procedure: adjuvant therapy
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) together with radiation therapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well surgery followed by gemcitabine, cisplatin, and radiation therapy works in treating patients with stage II or stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess overall survival and progression-free survival of patients with stage II-IIIB non-small cell lung cancer undergoing surgical resection, followed by adjuvant chemotherapy comprising gemcitabine and cisplatin, and radiotherapy.
* To assess the toxicities of this regimen in these patients.
* To evaluate the mRNA expression of enzymes (i.e., excision repair cross complementing protein, ribonucleotide reductase, and cytidine/deoxycytidine deaminase and kinase), which may be important in regulating the cytotoxicity of gemcitabine and cisplatin in patient tumors.
* To correlate mRNA levels with progression-free survival of patients treated with this regimen.
* To assess BCL2, P53, and HER2-neu expression by IHC and correlation with progression-free survival.

OUTLINE: Patients undergo surgical resection of their tumor and mediastinal lymph node dissection. Patients with complete surgical eradication of their disease or pathologic evidence of microscopic residual disease proceed to adjuvant chemotherapy.

Within approximately 60 days after surgical resection, patients receive adjuvant chemotherapy comprising gemcitabine IV over 30 minutes on days 1 and 8 and cisplatin IV over 1 hour on day 8. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

Beginning 130-144 days after surgery, patients undergo radiotherapy once daily, five days a week, for approximately 6 weeks.

Tumor tissue specimens are obtained at the time of surgical resection for pharmacodynamic and biomarker correlative studies. Specimens are examined by reverse transcriptase-polymerase chain reaction to measure mRNA expression of target oncogenes (i.e., DNA repair gene ERCC-1 and M2 subunit of the DNA repair gene ribonucleotide reductase) and enzymes (i.e., cytidine/deoxycytidine deaminase and kinase). Resected specimens are also assessed by IHC for the expression of BCL2, P53, and HER2-neu genes.

After completion of study therapy, patients are followed every 6 months for 5 years and annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed single, primary bronchogenic non-small cell lung cancer meeting the following subtypes:

  * Adenocarcinoma (no bronchioalveolar cell histology)
  * Squamous cell carcinoma
  * Large cell carcinoma
* Meeting the following staging criteria:

  * Stage IIB (T2, N1, M0, or T3, N0, M0)
  * Stage IIIA (T1-3, N2, M0 or T3, N1, M0)
  * Stage IIIB (Any T, N3, M0 or T4, Any N, M0)
* No more than 1 parenchymal lesion in the same lung or in both lungs
* No tumor involving the superior sulcus (e.g., Pancoast tumor)
* Patients must undergo evaluation by the involved thoracic surgeon, medical oncologist, and radiation oncologist prior to registration
* No evidence of metastatic disease

  * Biopsy or aspiration cytology required to confirm the benign diagnosis of CT or MRI abnormalities that potentially represent metastatic disease
  * Biopsy required if all noninvasive tests are indeterminant

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Absolute granulocyte count ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Bilirubin ≤ 3 times upper limit of normal (ULN)
* SGOT and SGPT ≤ 3 times ULN
* Creatinine clearance > 50 mL/min
* No prior malignancy except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, ductal or lobular carcinoma in situ of the breast, or any other cancer from which the patient has been disease-free for 5 years
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective protection
* No significant hearing loss or patient unwilling to accept potential for further hearing loss
* No uncontrolled medical illness by appropriate medical therapy (e.g., myocardial infarction within the past 3 months or liver cirrhosis)
* No symptomatic peripheral neuropathy affecting activities of daily living

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy for lung cancer

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 1999-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianna Koczywas, MD, Principal Investigator — City of Hope Comprehensive Cancer Center

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gemcitabine + Cisplatin
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 66 [63 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Two-year Progression-free Survival From the Date of Surgery
Description: Estimated using the product-limit method of Kaplan and Meier. Progression defined as a 25% increase or an increase of 10 cm2 (whichever is smaller) in the sum of the products of all measurable lesions over the smallest sum observed (over baseline if no decrease) using the same techniques as baseline, or clear worsening of any evaluable disease, or reappearance of any lesion that had disappeared, or appearance of any new lesion/site, or failure to return for evaluation or death, or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: 2 years post-surgery
Population: Study was terminated after accruing only three patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 3
percentage of participants | 67.6 [9.0 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

ADVERSE EVENTS:
Time Frame: Adverse events were recorded over a period of 46 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Gemcitabine + Cisplatin
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine + Cisplatin (N=3)
Hemoglobin decreased (Blood and lymphatic system disorders) | 3 (10)
Lymphangiopathy NOS (Blood and lymphatic system disorders) | 1 (1)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (1)
Packed red blood cell transfusion (Blood and lymphatic system disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (3)
Eye disorder (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (7)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (5)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (5)
Fever (General disorders) | 2 (2)
General symptom (General disorders) | 1 (1)
Oedema NOS (General disorders) | 1 (1)
Pain (General disorders) | 3 (9)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (3)
Creatinine increased (Investigations) | 2 (6)
Leukopenia (Investigations) | 2 (5)
Lymphopenia (Investigations) | 1 (3)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 1 (3)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 3 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (5)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (4)
Hyponatremia (Metabolism and nutrition disorders) | 1 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Taste alteration (Nervous system disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (2)
Hypotension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was closed early due to poor accrual. Reported data are not statistically powered to provide meaningful conclusions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes